## **PROVESA** trial

Proficiency based progression training for robotic vesico-urethral anastomosis chicken model versus the Halsted's model: a cross-specialty, multicentric, randomized and blinded clinical trial.

## **Informed Consent Form**

Principal Investigator: Ruben De Groote, MD

Research center: ORSI Academy, Melle, Belgium

July 27th 2020

NCT ID not yet assigned

Ethical Committee approval number 22072020

## DECLARATION OF THE PARTICIPANT IN THE STUDY

| Undersigned, |
|---|
| (name of the participant). |
| Hereby confirms that he/she has been informed about the nature, the characteristics, the duration and the purposes of the study. |
| Confirms to have received the information prior and in a timely fashion and gives permission to use the data collected. |
| Declares to be aware that the investigator may use his/her data, including previous surgical experiences state of education and training, video materials made during the performance of the exercises involved in the study, and all the other data in agreement with article 43 Code of the medical doctrine of duties for scientific purposes on condition that the publications do not mention any names or details that can make the identification of the participants by a third party possible, statistical processes, statistical analyses and may share anonimized data with third parties, on the basis of article 44 Code Code of the medical doctrine or duties, with the purpose of scientific research and/or publications under the supervision of the investigator |
| Confirms to have knowledge of the processing of personal data, the transmission of anonimized data to a third party with a view to scientific research, the rights of the involved and the complaint procedure as described in the privacy policy of the OLV Hospital Aalst, at which the previously mentioned has the qualification of the responsible for processing and has taken technical, organisatorical measures to guarantee the safety and integrity of the processed personal data. |
| Executed at (place) on (date) |
| (signature of the participant preceded by "read and approved") |